CLINICAL TRIAL: NCT06903455
Title: Effects of a Culturally Significant Cardiovascular Dance-based Intervention in Obese Women
Brief Title: A Culturally Significant Cardiovascular Dance-based Intervention in Obese Women
Acronym: CC-Dance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Catolica Silva Henriquez (Other)
Collaborators: Universidad Arturo Prat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FONDEPORTE; n°2400120062; n°2400120062 (Other Grant/Funding Number: FONDEPORTE, Instituto Nacional del Deporte (IND-Chile))
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Overweight, Obesity, Noncomunicable Diseases
Keywords: overweight, obesity, non-communicable diseases, exercise
MeSH Terms: conditions — Overweight; Obesity; Noncommunicable Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- culturally relevant cardio dance called Fitfolk (Experimental): "Fitfolk" is a new cardiovascular dance discipline that combines fitness exercises with music and dance from Chilean and Latin American folklore. This discipline promotes physical and emotional well-being and celebrates national folklore.
  Interventions: Other: Fit-folk cardio dance
- conventional physical exercise (Active Comparator): physical exercise program that contains resistance exercise and cardiorespiratory training
  Interventions: Other: Conventional physical exercise

INTERVENTIONS:
Other: Fit-folk cardio dance — "Fitfolk" is a new cardiovascular dance discipline that combines fitness exercises with music and dance from Chilean and Latin American folklore. This discipline promotes physical and emotional well-being and celebrates national folklore.
  Arms: culturally relevant cardio dance called Fitfolk
Other: Conventional physical exercise — conventional physical exercise program that uses resistance exercise and cardiorespiratory training
  Arms: conventional physical exercise

SUMMARY:
The objective of this study is to analyze a culturally relevant cardiovascular dance-based intervention called Fitfolk in overweight or obese Mapuche women from a rural community in Padre las Casas. Participants will be randomly assigned to two groups: an experimental group that will receive a culturally relevant cardiovascular dance program (EG, n=11), and a control group that will receive a conventional physical exercise program (CG, n=11). Both groups will be trained at a community center in the same rural area, led by a physical education professional. The principle of training progression will be followed, and they will exercise three times per week with sessions of approximately one hour for 12 weeks. Physical health parameters, quality of life, motivation, and barriers to physical exercise will be assessed.

DETAILED DESCRIPTION:
Design: A two-arm randomized controlled trial conducted according to the CONSORT declaration. The design considers single blinding. The protocol will be based on the Singapore Declaration, and all participants must voluntarily sign a consent form. The protocol will be submitted to the Scientific Ethics Committee of the Araucanía Sur Health Service.

Sample: The sample will consist of 22 adult women from rural areas of the Padre las Casas commune. The sample will be selected using a non-probability convenience method, with those who meet the inclusion criteria: women aged ≥18 years, sedentary according to WHO criteria, diagnosed with excess malnutrition (overweight/obesity), and with controlled chronic diseases (diabetes, hypertension, dyslipidemia). Those with organic pathologies that preclude physical activity, such as stroke, myocardial infarction, neurological diseases, or uncontrolled chronic diseases, will be excluded. Participants will be randomly assigned to two groups. An experimental group will receive a culturally relevant cardiovascular dance program (EG, n=11) and a control group will receive a conventional physical exercise program (CG, n=11). Both groups will receive exercise at locations in the same rural areas, led by a physical education professional. The principle of training progression will be followed, and they will exercise three times per week with sessions of approximately one hour for 12 weeks.

Procedures: An agreement will be established with two communities in rural areas of Padre las Casas, with an initial contact between an anthropologist and community leaders. The lead researcher will contact potential participants to inform them about the characteristics of the research and request their informed consent.

Instruments and variables: Assessments will be conducted before and after each intervention.

a. Physical health: Handgrip strength with dynamometry, cardiovascular endurance with the Shuttle walking test, flexibility with the Sit and Reach test, blood pressure with a sphygmomanometer, glycosylated hemoglobin (HbA1c) with a blood test, lipid profile with a blood test, anthropometry (weight, height, weight, waist-hip ratio), physical activity with the Basic Physical Activity Questionnaire (GPAQ),

a. Quality of life: with the quality of life questionnaire (SF-36).

a. Motivation and Barriers to exercise: Motivation for physical exercise with the Exercise Behavior Regulation Questionnaire (BREQ-3), and barriers and physical benefits to physical exercise with the Exercise Benefits/Barriers Scale (EBBS).

In addition, sociodemographic data will be collected, and control variables will be measured before, during, and after each exercise session.

Statistical analysis: The sample size was calculated a priori using G*Power 3.1.9.7. Sixteen subjects in total were required (8 in each group) considering α=0.05, 1-β=0.8 and effect size (ES)=1.32 for aerobic capacity based on the results of a previous study. Considering the possibility of dropout, 6 subjects were added (total n=22; n=11 in each group). The description will be done as measures of central tendency and dispersion (continuous variables) and as percentages (categorical variables). The Shapiro-Wilk test will be used to verify the normality of the data. A two-way repeated measures analysis of variance (ANOVA) will be used to determine the effects of the interventions. The Bonferroni post hoc test will be applied to identify statistically significant comparisons. All analyses will be performed using SPSS v.25 (SPSS, Inc., Chicago, IL, USA) considering p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old,
* Belonging to the Huichacura-Cayuqueo indigenous community.
* Sedentary, according to WHO criteria.
* Diagnosed with malnutrition due to excess (overweight/obesity).
* With controlled chronic diseases (diabetes, hypertension, dyslipidemia).

Exclusion Criteria:

-Those with organic pathologies that make it impossible to engage in physical activity, such as stroke, myocardial infarction, neurological diseases, or uncontrolled chronic diseases, will be excluded.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Improvement in the physical condition of the participants related to the intervention, according to the ST3x1 step test | from the start of treatment until its completion at 12 weeks
  Its best measurement is maximum oxygen consumption, which will be measured using the ST3x1 step test. assessed as relative vo2max (mL/kg/min), where higher values indicate improvements in cardiorespiratory fitness.
Improvements in participants' physical strength related to the intervention | From the start of treatment to its completion at 12 weeks
  Physical strength will be assessed using the 5-times sit-to-stand test and handgrip dynamometry. A decrease in the time spent sitting and standing 5 times and an increase in hand grip in kilograms will indicate an increase in physical strength.
Improvement in participants' long-term glycemic control relative to the intervention, as measured by glycated hemoglobin assay | from the start of treatment until its completion at 12 weeks
  This variable will be measured by a blood test that measures the average blood glucose level over the last two or three months, the result is presented as a percentage.

SECONDARY OUTCOMES:
Improvement in participants' quality of life in relation to the intervention, according to the WHOQOL-BREF quality of life questionnaire | from the start of treatment until its completion at 12 weeks
  The Woqhol-Bref Quality of Life Scale is a self-report questionnaire that assesses quality of life in four domains: physical health, psychological health, social relationships, and environment. Each domain is scored on a transformed scale from 0 to 100, with lower scores indicating poorer quality of life and higher scores indicating better quality of life.
Improvement in participants' physical activity compared to the intervention, according to the International Physical Activity Questionnaire (IPAQ). | from the start of treatment until its completion at 12 weeks
  The International Physical Activity Questionnaire (IPAQ) assesses physical activity levels using questions covering four domains: activity at work, at home, during transportation, and in leisure time. IPAQ results are expressed in MET-minutes per week (MET-min/wk), with higher values indicating higher levels of physical activity. Participants are also classified into three categories according to their physical activity level: low, moderate, and high.
Improvement in participants' motivation to engage in physical activity relative to the intervention, according to the "BREQ-3" exercise behavior regulation questionnaire. | from the start of treatment until its completion at 12 weeks
  The Exercise Behavior Regulation Questionnaire (BREQ-3) is a 23-item self-report instrument designed to assess different forms of motivational regulation toward physical exercise, based on the principles of Self-Determination Theory. The questionnaire is structured into six factors: intrinsic motivation, integrated regulation, identified regulation, introjected regulation, external regulation, and amotivation.
  Each item is answered on a 5-point Likert-type scale, ranging from 0 ("not at all true for me") to 4 ("very true for me"). Higher scores on the more self-determined regulation factors (such as intrinsic, integrated, and identified motivation) indicate more favorable motivation toward exercise, while high scores on external regulation or amotivation reflect less autonomous or unfavorable motivation.
Improvements in perceived barriers and benefits to physical exercise among participants in relation to the intervention, according to the Exercise Benefits and Barriers Scale (EBBS). | from the start of treatment until its completion at 12 weekS
  The perception of benefits and barriers to physical activity will be assessed using the Exercise Benefits and Barriers Scale (EBBS). This instrument consists of 43 items divided into two subscales: one assessing perceived benefits (29 items) and another measuring perceived barriers (14 items). Each item is answered using a 4-point Likert-type scale, ranging from 1 ("strongly disagree") to 4 ("strongly agree").
  Higher scores on the benefits subscale indicate a more positive perception of physical activity, while higher scores on the barriers subscale reflect greater perceptions of obstacles to physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Comunidad indigena Huichacura Cayuqueo, Padre Las Casas, Región de la Araucanía, Chile

IPD SHARING:
Plan to Share IPD: No